CLINICAL TRIAL: NCT01657656
Title: Vitamin D Supplementations as Adjunct to Anti-Tuberculosis Drugs in Mongolia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Ganmaa Davaasambuu, Assistant Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R00HL089710 (NIH)
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Vitamin D Supplements; Tuberculosis; Sputum; Cytokines; Immunity
MeSH Terms: conditions — Tuberculosis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D group (Experimental): Vitamin D supplement by Tishcon
  Interventions: Dietary Supplement: Vitamin D
- Control group (Placebo Comparator): Identically appearing capsules
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D

SUMMARY:
Hypothesis

That improving vitamin D status among TB patients will speed the pace of bacteriological cure, and will enhance immune responses to TB infection

DETAILED DESCRIPTION:
Tuberculosis (TB) will be the world's largest single cause of death from infection for the 30-year period between 1990 and 2020. More than 95% of TB cases, and deaths due to TB, occur in developing countries. Mongolia is one of the countries with the highest tuberculosis burdens in the Western Pacific region. In addition, vitamin D deficiency is endemic in Mongolia. We propose to determine the efficacy of vitamin D supplements, as an adjunct to multidrug therapy, in enhancing the anti-microbial immune response to TB, a finding that could lead to the development of shorter drug regimens, and thus more efficient and effective TB treatment protocols.

We propose to conduct a double blind, placebo controlled, randomized clinical trial to test the effect of a daily vitamin D supplementation on the ability of subjects to control TB infection.

The Primary Endpoint: The primary endpoint will be: time to sputum culture conversion from positive to negative. The number of days to sputum conversion will be measured, in both the intervention and control groups, starting on the date that treatment is begun. Sputum samples will be collected and cultured every two weeks thereafter. The date of conversion from positive to negative, for each subject, will be the date halfway between the date of the last culture-positive sputum and the first culture-negative one.

Secondary Endpoints:

Bacteriologic secondary endpoints, cell-mediated immune function endpoints and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Sputum positive TB patients

Exclusion Criteria:

* We will exclude those with abnormal LFTs at baseline (2.5 times upper limit of normal), as they will be at higher risk of developing drug-induced hepatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be time to sputum culture conversion from positive to negative. | Eight weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Communicable Dieases, Ulaanbaatar, Mongolia

REFERENCES:
- [Derived] Ganmaa D, Munkhzul B, Fawzi W, Spiegelman D, Willett WC, Bayasgalan P, Baasansuren E, Buyankhishig B, Oyun-Erdene S, Jolliffe DA, Xenakis T, Bromage S, Bloom BR, Martineau AR. High-Dose Vitamin D3 during Tuberculosis Treatment in Mongolia. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2017 Sep 1;196(5):628-637. doi: 10.1164/rccm.201705-0936OC. PMID 28692301